CLINICAL TRIAL: NCT03134391
Title: Comparison Between Vapocoolant Spray and Eutectic Mixture of Local Anesthetics in Reducing Pain From Spinal Injection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Riyadh Firdaus, Anesthesiologist Consultant, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: IndonesiaUAnes012
Record Dates: First submitted 2017-04-25; First posted 2017-05-01 (Actual); Last update posted 2017-08-18 (Actual); Status verified 2017-08

CONDITIONS: Adult Patient Undergoing Elective Surgery With Spinal Anesthesia
MeSH Terms: interventions — Lidocaine, Prilocaine Drug Combination

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- vapocoolant spray (Active Comparator): Subjects received Vapocoolant spray before spinal anesthesia
  Interventions: Drug: Vapocoolant spray, EMLA
- EMLA (Active Comparator): Subjects received EMLA before spinal anesthesia
  Interventions: Drug: Vapocoolant spray, EMLA

INTERVENTIONS:
Drug: Vapocoolant spray, EMLA — Subjects were given vapocoolant spray to reduce pain from spinal injection; subjects were given EMLA to reduce pain from spinal injection

SUMMARY:
This study aimed to evaluate the effect of vapocoolant spray and EMLA in reducing pain from spinal injection

DETAILED DESCRIPTION:
Approval from Ethical Committee of Faculty of Medicine Universitas Indonesia was acquired prior conducting the study. Subjects were given informed consent before enrolling the study and randomized into two groups (Vapocoolant spray group and eutectic mixture local anesthetics (EMLA) group). Intravenous (IV) cannulae with Ringer Acetate fluid, non-invasive blood pressure monitor, and pulse-oxymetry were set on the subjects in the operation room. Vital signs were recorded. Patients were positioned in sitting position and were instructed to flex their head and bend their back. Identification of intervertebral space L4-5 were performed. Asepsis and antisepsis procedure were performed. The Vapocoolant spray group received vapocoolant spray at a distance of 10 cm for 2 seconds and we waited for 10 seconds. The EMLA group received EMLA cream which consisted of 2.5% lidocaine and 2.5 % prilocaine in 2 ml of water/oil emulsion and then they received tegaderm as the dressing for 45-60 minutes before the cream was wiped off. Spinal injection using 27G needle were performed after the intervention to each groups. Needle bevels were aligned parallel to dura fibres. Patients' visual analog score (VAS) and movements were recorded. Evaluation was only done in the first injection attempt, and was followed until the depth of the needle was around 5 mm. After the injection was successfully performed, patients' position were changed into supine position. Evaluation and recording were performed by person who was blinded from the intervention. Vital signs were recorded for every 3 minutes in the first 15 minutes, and then every 5 minutes until the end of the procedure.

ELIGIBILITY:
Inclusion Criteria:

* woman aged >18 years old
* American Society of Anesthesiologists (ASA) physical status I-III who were planned to undergo one-day care elective surgery at operating room in spinal anesthesia
* patients who were planned to undergo brachytherapy

Exclusion Criteria:

* Subjects with history of allergy to anesthetic agents
* unstable hemodynamic
* history of active psychotropic drug consumption
* spinal anesthesia contraindications such as local infection, severe coagulopathy, severe hypovolemia, or increased intracranial pressure

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Studies has shown that women have lower threshold for pain
Enrollment: 97 (Actual)
Dates: Start 2016-08-01 (Actual); Primary Completion 2016-10-30 (Actual); Study Completion 2017-05-31 (Actual)

PRIMARY OUTCOMES:
VAS | Day 1
  Visual Analog Scale for measuring pain
Vital signs | day 1
  Vital signs for measuring pain indirectly

CONTACTS AND LOCATIONS:
Locations (1):
- Cipto Mangunkusumo Cental National Hospital, Jakarta, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bujedo BM. Current evidence for spinal opioid selection in postoperative pain. Korean J Pain. 2014 Jul;27(3):200-9. doi: 10.3344/kjp.2014.27.3.200. Epub 2014 Jun 30. PMID 25031805
- [Background] Bujedo BM, Santos SG, Azpiazu AU. A review of epidural and intrathecal opioids used in the management of postoperative pain. J Opioid Manag. 2012 May-Jun;8(3):177-92. doi: 10.5055/jom.2012.0114. PMID 22798178
- [Result] Kim SH, Jeon DH, Chang CH, Lee SJ, Shin YS. Spinal anesthesia with isobaric tetracaine in patients with previous lumbar spinal surgery. Yonsei Med J. 2009 Apr 30;50(2):252-6. doi: 10.3349/ymj.2009.50.2.252. PMID 19430559
- See also: Kim YJ, Jung MH, Choi YR, Park HJ, Won RS, Lee JY, et al. The analgesic efficacy of a 5% eutectic mixture of lidocaine and prilocaine prior to insertion of spinal and epidural block. Korean J of Anesthesiol. 2008;54(4):395-9. — https://synapse.koreamed.org/DOIx.php?id=10.4097/kjae.2008.54.4.395&vmode=PUBREADER